CLINICAL TRIAL: NCT05318326
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Trial to Evaluate the Clinical Efficacy and Safety of Yogliptin Tablets in Chinese Patients With Type 2 Diabetes Mellitus and Poor Diet and Exercise Control
Brief Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Trial to Evaluate the Clinical Efficacy and Safety of Yogliptin Tablets
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengdu Easton Biopharmaceuticals Co,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ChengduEastonBiopharma
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo control group (Placebo Comparator): Placebo control group
  Interventions: Drug: placebo group
- Yogliptin 200mg group (Experimental): Yogliptin 200mg group
  Interventions: Drug: Yogliptin 400mg group
- Yogliptin 400mg group (Experimental): Yogliptin 400mg group
  Interventions: Drug: Yogliptin 200mg group

INTERVENTIONS:
Drug: placebo group — placebo 400mg (4 tablet) , Q1W, oral, week 1 to week 24; Yogliptin 400 mg (4 tablet), Q1W, oral, week 25 to week 52.
  Arms: Placebo control group
Drug: Yogliptin 400mg group — Yogliptin 400mg (4 tablet) , Q1W, oral, week 1 to week 24; Yogliptin 400 mg (4 tablet), Q1W, oral, week 25 to week 52.
  Arms: Yogliptin 200mg group
Drug: Yogliptin 200mg group — Yogliptin 200mg (2 tablet) and placebo 200 mg (2 tablet), Q1W, oral, week 1 to week 24; Yogliptin 400 mg (4 tablet), Q1W, oral, week 25 to week 52.
  Arms: Yogliptin 400mg group

SUMMARY:
The purpose of this study is to assess the efficacy of Yogliptin (as monotherapy) compared with placebo after 24 weeks, and the safety (up to 52 weeks) of Yogliptin in Chinese patients with Type 2 diabetes who are insufficient glycaemic control with diet and exercise.

DETAILED DESCRIPTION:
The treatment period is composed of a 24-week double-blind period (week 1-24) and a 28-week open-label period (week 25-52). During the double-blind period, participants will receive 200 mg or 400 mg dose of Yogliptin and matching placebo, or placebo only. During the open-label period, all participants will receive 400 mg dose of Yogliptin.

ELIGIBILITY:
Inclusion Criteria:

* 1.Men or women aged 18 to 75 years old at the day of signing the informed consent;
* 2.Type 2 diabetes patients who meet the diagnostic criteria for diabetes issued byChinese Guidelines for the Prevention and Treatment of Type 2 Diabetesin 2020;
* 3.Receive at least 8 weeks of diet and exercise treatment before screening;Not treated with any antidiabetic drugs within 8 weeks before screening;
* 4.Glycated hemoglobin (HbA1c): Screening period: HbA1c 7.5% to 11% (tested by the research center), when randomly enrolled: HbA1c 7.0% to 10.5% (central laboratory test) Measurement);

  5.fasting blood glucose(FPG): Screening period: FPG≤15.0mmol/L (tested by the research center), when randomly enrolled: FPG≤15.0mmol/L (central laboratory test) Measurement);
* 6.Screening period Body mass index(BMI) 19.0kg/m2 to 35.0kg/m2 ;
* 7.Agree to maintain the same diet and exercise habits throughout the trial and be willing and able to accurately use a home blood glucose meter for self-monitoring and recording of blood glucose
* 8.Can understand the procedures and methods of this study, willing to strictly abide by the clinical trial protocol to complete this trial, and voluntarily sign an informed consent.

Exclusion Criteria:

* 1.Non-type 2 diabetes: such as type 1 diabetes, secondary diabetes or other special types of diabetes ；
* 2.History or condition of any of the following at screening or run-in:Those who have a history of diabetic ketoacidosis, hyperglycemia and hyperosmolarity, lactic acidosis and other acute complications of diabetes within 6 months before screening;
* 3.History or condition of any of the following at screening or run-in:Unstable condition or severe diabetic complications such as proliferative retinopathy or maculopathy, severe diabetic neuropathy, intermittent claudication, diabetic foot in the past 6 months；
* 4.History or condition of any of the following at screening or run-in:Three or more episodes of grade 3 hypoglycemia in the past 6 months (according to the diagnostic criteria for hypoglycemia in the Chinese Guidelines for the Prevention and Treatment of Type 2 Diabetes (2020 edition)) ;
* 5.History or condition of any of the following at screening or run-in:Unstable angina, stroke or transient ischemic attack, myocardial infarction, coronary artery bypass graft or percutaneous coronary intervention (diagnostic angiography is allowed of);
* 6.History or condition of any of the following at screening or run-in:Hemorrhagic stroke or ischemic stroke within the past 6 months, and is not suitable for this clinical trial judged by the investigator ;
* 7. History or condition of any of the following at screening or run-in:Previous history of other serious endocrine diseases affecting glucose metabolism, such as multiple endocrine neoplasia, limb hypertrophy syndrome, Cushing's syndrome, etc., which are not suitable for this clinical trial judged by the ;
* 8. History or condition of any of the following at screening or run-in:Patients with previous severe digestive system diseases, nutritional metabolic diseases and rheumatic diseases, who are not suitable to participate in this clinical trial as judged by the investigator；
* 9. any of the following medical history or conditions at screening or run-in: current thyroid dysfunction not controlled with stable drug dose, and clinically significant abnormalities in thyroid function test results at screening
* 10 Any of the following medical history or conditions at screening or run-in: History or presence of malignancy (except for malignancies that have not recurred in the last 5 years)
* 11 History or condition of any of the following at screening or run-in: Presence of significant psychiatric disorder or speech disorder Unwilling or unable to fully understand and collaborate Contacts and Locations
* 12 Any of the following medical history or conditions at screening or run-in: significant infection or major surgery within 6 months prior to screening, which, in the judgment of the investigator, would make the patient inappropriate for this clinical trial ;
* 13 History or conditions of any of the following at screening or run-in: those with a history or clinical evidence of acute or chronic pancreatitis；
* 14 History or condition of any of the following at screening or run-in: poorly controlled blood pressure, ie, systolic blood pressure (SBP) > 160 mmHg and/or diastolic blood pressure (DBP) > 100 mmHg ;
* 15 Use of any of the following medications or therapies prior to Screening or Run-in: Dipeptidyl peptidase-4 (DPP-4) inhibitors, glucagon-like peptide-1 (GLP-1) receptor agonists prior to Screening or within 3 months prior to Run-in ;
* 16 Use of any of the following drugs or therapies before screening or run-in: Use of other drugs that may affect glucose metabolism, such as systemic glucocorticoids, growth hormone, etc., before screening or within 3 months before run-in;
* 17 Use of any of the following drugs or therapies before screening or run-in: those with cumulative use of insulin and its analogues for more than 28 days in the previous year (except for gestational diabetes treated with insulin and its analogues)
* 18. When screening, any one of the laboratory inspection indicators meets the following standards: ALT/AST> 2.5ULN; Total bilirubin> 2.0ULN; Subjects with current severe renal disease, or eGFR (CKD-EPI2012Scr-CysC) ≤ 60 mL/min/1.73 m2;TG）>5.6mmol/L;Blood amylase>>1.5ULN;HGB<10.0g/dL（100g/L）;
* 19 Any positive HCV antibody, HIV antibody or Treponema pallidum antibody at screening; positive hepatitis B HBsAg, additionally test hepatitis B virus load (HBV-DNA), positive HBsAg and HBV-DNA higher than the lower limit of detection in the local laboratory;
* 20 .The patient may have any contraindications, allergies or hypersensitivity to Test drug (including study drug and placebo) or its excipients, DPP4 drugs
* 21.Patients with a history of joint pain after taking DPP-4 inhibitors ;
* 22.Patients who have received 3 or more times of clinical trial drugs within the past year, or patients who have received 1 time of clinical trial drugs within 1 month before screening ;
* 23 Female subjects who are pregnant, lactating, or planning pregnancy during the study ;
* 24 Male and female subjects of childbearing potential who do not agree to practice contraception during the study. Females of childbearing potential (including those less than 2 years postmenopausal) must agree to practice a reliable method of contraception (e.g., transdermal contraceptive patch, implantable long-acting solution for injection, contraceptive ring, subdermal implant, intrauterine device, or double barrier method (diaphragm+condom) throughout the entire study period) ;
* 25 One or more grade 3 hypoglycemic events without obvious cause during the run-in period ；
* 26 Medication compliance with the lozenge was < 75% or > 125% during the run-in period ；
* 27 The subject has any other factors that the investigator considers inappropriate for the trial 。

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c change from baseline at week 24 | Baseline and week 24
  Change From Baseline in Hemoglobin A1c (HbA1c) at Week 24

SECONDARY OUTCOMES:
FPG Change From Baseline at Week 24 and Week 52 | Baseline, week 24 and week 52
2h-PPG Change From Baseline at Week 24 and Week 44 and Week 52 | Baseline, week 24 and Week 44 and Week 52
Percentage of Patients With HbA1c <6.5% | Time Frame: Baseline, week 24 and week 52
Percentage of Patients With HbA1c <7.0% | Baseline, week 24 and week 52
blood pressure Change From Baseline at Week 24 and Week 52 | Baseline, week 24 and week 52
Weight Change From Baseline at Week 24 and Week 52 | Baseline, week 24 and week 52
Fasting lipids From Baseline at Week 24 and Week 52 | Baseline, week 24 and week 52

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Guo, Study Director — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China